CLINICAL TRIAL: NCT05946343
Title: The Relationship Between Rotator Cuff Tear Severity and Scapular and Rotator Cuff Muscle Activation Patterns: A Cross-Sectional Study
Brief Title: Rotator Cuff Tear Severity and Scapular and Rotator Cuff Muscle Activation Patterns
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Other Study IDs: 012/09978882023
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Injuries; Shoulder Pain
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain | interventions — Electromyography; Physical Examination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Small Rotator Cuff Tear Group: The Cofield classification system is a commonly cited classification system for full-thickness rotator cuff tears. It is based on the size of the tear. Small tear: Less than 1 cm.
  Interventions: Diagnostic Test: Surface Electromyography (sEMG) Assessment
- Medium Rotator Cuff Tear Group: The Cofield classification system is a commonly cited classification system for full-thickness rotator cuff tears. It is based on the size of the tear. Medium tear: 1-3 cm
  Interventions: Diagnostic Test: Surface Electromyography (sEMG) Assessment
- Large Rotator Cuff Tear Group: The Cofield classification system is a commonly cited classification system for full-thickness rotator cuff tears. It is based on the size of the tear. Large tear: 3-5 cm
  Interventions: Diagnostic Test: Surface Electromyography (sEMG) Assessment
- Massive Rotator Cuff Tear Group: The Cofield classification system is a commonly cited classification system for full-thickness rotator cuff tears. It is based on the size of the tear. Massive tear: Greater than 5 cm
  Interventions: Diagnostic Test: Surface Electromyography (sEMG) Assessment

INTERVENTIONS:
Diagnostic Test: Surface Electromyography (sEMG) Assessment — Surface electromyography (sEMG) will be used to assess the activation patterns of scapular and rotator cuff muscles during functional tasks, such as shoulder flexion, abduction, and external rotation. The sEMG assessment will be conducted using a wireless sEMG system with a sampling rate of 2000 Hz and a bandwidth of 20-500 Hz. Pre-gelled, disposable, self-adhesive Ag/AgCl electrodes will be placed on the muscle belly according to SENIAM guidelines, with an inter-electrode distance of 20 mm.

SUMMARY:
Rotator cuff tears are common musculoskeletal injuries that can lead to altered scapular and rotator cuff muscle activation patterns and reduced function. This study aims to investigate the relationship between rotator cuff tear severity and scapular and rotator cuff muscle activation patterns.

The primary objective of this study is to determine whether a relationship exists between the severity of rotator cuff tears and the activation patterns of scapular and rotator cuff muscles. Secondary objectives include:

1. Identifying differences in muscle activation patterns between varying tear sizes.
2. Evaluating the potential of these activation patterns as an indicator for the severity of rotator cuff tears.
3. Assessing the influence of muscle activation patterns on the functional capacity of the affected shoulder.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years.
* Diagnosis of rotator cuff tear confirmed by a qualified orthopedic surgeon.
* MRI scan showing the size of the tear (small, medium, large, or massive).
* Ability to provide informed consent and comply with the study protocol.

Exclusion Criteria:

* History of shoulder surgery or other shoulder disorders unrelated to rotator cuff tears.
* Presence of neurological, cardiovascular, or respiratory disorders that could influence muscle activation patterns.
* Contraindications for sEMG assessment, such as skin allergies or infections.
* Inability to perform the required functional tasks due to severe pain or disability.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population for this research will be individuals between the ages of 18-60 years with a diagnosis of rotator cuff tears confirmed by magnetic resonance imaging (MRI). Participants will be recruited from orthopaedics and hospitals in the local area.
  Participants will be stratified based on tear size (small, medium, large, or massive) as determined by MRI.
  Participants will be fully informed of the objectives, procedures, potential risks, and benefits of the study, as well as their right to withdraw from the study at any time without penalty. Informed consent will be obtained from all participants prior to their enrolment in the study.
  The study population will be diverse in terms of age, sex, tear size, and symptom severity, which will enable the findings to be generalized to a broader population with rotator cuff tears.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Muscle Activation Amplitude | baseline
  Muscle activation amplitude for the scapular and rotator cuff muscles (serratus anterior, upper and lower trapezius, supraspinatus, and infraspinatus) during functional tasks.

SECONDARY OUTCOMES:
Differences in Muscle Activation Patterns by Tear Size | baseline
  Identification of differences in muscle activation patterns between varying tear sizes (small, medium, large, and massive).

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Chair — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No